CLINICAL TRIAL: NCT06708585
Title: Effects of Planned Pre-Cesarean Information and Progressive Relaxation Exercises on Surgical Fear, Anxiety, Postpartum Comfort and Pain Levels of Primigravida Women: A Randomized Controlled Trial
Brief Title: Information and Progressive Relaxation Exercises
Acronym: RKÇ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIGDE OMER HALISDEMIR UNIVERSI
Record Dates: First submitted 2024-09-24; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-09

CONDITIONS: Caesarean Section; Fear; Anxiety; Pain
Keywords: Cesarean section, fear, anxiety, comfort, pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: The research is a two-group parallel randomized controlled experimental study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Each pregnant woman who meets the inclusion criteria will be interviewed individually for approximately 15-20 minutes on the day of surgery and data collection forms will be applied. Then, each woman will be given progressive relaxation exercises individually. Exercises will begin two hours before surgery and will be repeated four times. Each exercise will last approximately 20 minutes. Data collection forms will be applied two hours after the completion of the exercise and at the end of surgery.
  Interventions: Other: progressive relaxation exercises and training
- control group (No Intervention): Each pregnant woman in the control group will be administered the individual information form, State Anxiety Scale, and Surgical Fear Scale data collection tools two hours before the surgery and will be released to the routine care of the institution. After two hours, the State Anxiety Scale and Surgical Fear Scale will be administered again. 6 hours after the cesarean section, the woman's pain will be assessed with the VAS pain scale and 24 hours later, the postpartum comfort scale will be administered.

INTERVENTIONS:
Other: progressive relaxation exercises and training — Considering the high incidence of cesarean section and the prevalence of anxiety and fear as psychological symptoms, providing comfort and pain support to women is of great importance. Therefore, the effect of progressive relaxation exercise and education before cesarean section surgery on care outcomes will be determined.
  Arms: Experimental group

SUMMARY:
This study was planned to determine the effect of information and progressive relaxation exercises before planned cesarean section on surgical fear, anxiety, postpartum comfort and pain levels.The research will be conducted in experimental design. The research will begin after receiving written permission from Niğde Ömer Halisdemir University Ethics Committee, Niğde Provincial Health Directorate and Ömer Halisdemir Training and Research Hospital. Pregnant women who are between the ages of 18-35, who are on Primigravida, who apply for a planned cesarean section, who have a live single pregnancy, and who are planned for spinal anesthesia will be included in the study. Before starting the research, the study will begin by obtaining institutional permissions and written permission from the pregnant women. Pre-Assessment Form, Personal Information Form, State Anxiety Scale, Surgical Fear Scale, Postpartum Comfort Scale will be used to collect data. The data will be evaluated on a computer using the IBM SPSS Statistics 24 (Statistical Package for the Social Sciences for Windows) package program. Appropriate statistical analyzes will be used to evaluate the data.

DETAILED DESCRIPTION:
There is an increase in the frequency of cesarean sections worldwide (Abdelrahman et al., 2020). WHO states that approximately 18.6 million cesarean sections are performed annually. It is observed that the frequency of cesarean sections in Turkey is increasing every year. According to the Health Statistics Yearbook 2021 data, the rate of cesarean sections in live births is 58.4%, and the rate of primary cesarean sections in live births is 29.1%. These rates show that they are well above the ideal cesarean rate determined by WHO, which should be between 10-15%.

Although there are many known reasons for the increase in cesarean sections, more than 80% of women experience fear and anxiety before and during cesarean sections (Abarghoee et al., 2022; Salmanzadeh et al., 2018). A significant portion of women who undergo cesarean sections experience high levels of anxiety before the procedure (Maleki et al., 2022). Studies show that 63-86% of women who undergo cesarean section have higher levels of fear and anxiety compared to those who undergo general surgery (Ferede et al., 2022). Anxiety related to cesarean section surgery has been associated with physiological and psychological risks. Fear and anxiety experienced before cesarean section can trigger responses from both the sympathetic and parasympathetic nervous systems, as well as affecting hormone levels. As a result, these responses can lead to increased blood pressure and heart rate, and cardiac arrhythmia (Koca et al. 2021). In addition, excessive fear and anxiety before and during surgery can lead to anesthesia complications, increased need for postoperative pain relief, prolonged recovery, delayed initiation of breastfeeding and discharge, higher costs, and decreased satisfaction with the birth experience (Schaal et al. ., 2020 and Hepp et al., 2018). Therefore, it is particularly important to address and reduce fear and anxiety related to cesarean section, as lower levels of fear and anxiety before and during surgery have been associated with greater maternal satisfaction and a more positive overall birth experience (Noben et al., 2019). Managing fear and anxiety can be approached using both pharmaceutical and non-pharmacological methods. Although pharmaceutical approaches are widely used, they can be expensive, sometimes painful, and carry the potential risk of adverse effects on the fetus if they cross the placenta (Eslami et al., 2020). Therefore, there is a focus on using non-pharmacological techniques to alleviate fear and anxiety in women undergoing cesarean section (Abadi et al., 2018). One effective example is the use of relaxation techniques to reduce fear and anxiety (Vagnoli et al., 2019). Frequently used methods include meditation, massage therapy, muscle relaxation exercises, acupuncture, energy healing applications, different breathing techniques such as controlled breathing or diaphragmatic breathing (Mohamady et al. 2022). Relaxation exercise is associated with decreased oxygen consumption levels and decreased activity in the sympathetic nervous system (Ibrahim et al., 2019). One of the known methods of achieving relaxation is progressive relaxation exercise (PGE). Technically, PGE involves the voluntary, systematic tension and complete relaxation of large muscle groups until relaxation is achieved throughout the body. The aim is to ensure that the individual can relax on their own in their daily lives by feeling the difference between tension and relaxation in their body and mind (Burke et al. 2011; Özveren 2011). Considering the high incidence of cesarean section and the prevalence of anxiety and fear as psychological symptoms, it is of great importance to provide comfort and pain support to women. Therefore, the aim of this study was to determine the effects of planned pre-cesarean information and progressive relaxation exercises on surgical fear, anxiety, postpartum comfort and pain levels of primiparous women.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-35,
* Primigravida,
* Applied for planned cesarean section,
* Live singleton pregnancy,
* Spinal anesthesia planned,

Exclusion Criteria:

* Women who develop postpartum maternal or neonatal complications
* Receiving general anesthesia.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — primigravida women
Enrollment: 68 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2025-02-20 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
State Anxiety Scale | 3 month
  It is understood that as the score obtained from the scale increases, anxiety increases.
Surgical Fear Scale | 3 month
  a high score indicates that surgical fear is high

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | 3 month
  It consists of a 10 cm long horizontal or vertical line, which is frequently used in the measurement of subjective parameters.
postpartum comfort scale | 3 month
  The lowest score that can be obtained from the scale is 34, while the highest score is 170.

CONTACTS AND LOCATIONS:
Overall Officials: birnur YEŞİLDAĞ, Dr, Study Director — Ömer Halisdemir University
Locations (1):
- Ömer Halisdemir University Training and Research Hospital, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No